CLINICAL TRIAL: NCT02246153
Title: Morbidity and Mortality of Laparoscopy-assisted and Open Distal Gastrectomy for Gastric Cancer in the Elderly Patients: A Randomized Controlled Trial
Brief Title: Laparoscopy-assisted and Open Distal Gastrectomy for Gastric Cancer in the Elderly Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Guoxin Li, M.D.,Ph.D., F.R.C.S., Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2014-067
Record Dates: First submitted 2014-09-15; First posted 2014-09-22 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Complications
Keywords: Laparoscopic gastrectomy; Advanced gastric cancer; Elderly patients; Morbidity; Mortality

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic gastrectomy (Experimental): Laparoscopy-assisted distal gastrectomy with D2 lymphadenectomy will be performed for the treatment of patients assigned to this group.
  Interventions: Procedure: Laparoscopic gastrectomy
- Open gastrectomy (Active Comparator): Open distal gastrectomy with D2 lymphadenectomy will be performed for the treatment of patients assigned to this group.
  Interventions: Procedure: Open gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic gastrectomy — * After exclusion of T4b, bulky lymph nodes, or distant metastasis case by diagnostic laparoscopy, laparoscopic distal subtotal gastrectomy and D2 lymph node dissection will be performed with curative treated intent.
  * The type of reconstruction will be selected according to the surgeon's experience and anastomotic procedure is performed extracorporeally using a mini-laparotomy.
  Other Names: LDG
  Arms: Laparoscopic gastrectomy
Procedure: Open gastrectomy — * After exclusion of T4b, bulky lymph nodes, or distant metastasis case by diagnostic laparoscopy, open distal subtotal gastrectomy and D2 lymph node dissection will be performed with curative treated intent.
  * The type of reconstruction will be selected according to the surgeon's experience.
  Other Names: ODG
  Arms: Open gastrectomy

SUMMARY:
* Laparoscopy-assisted distal gastrectomy for the treatment of early gastric cancer (EGC) has been supported by high-quality evidence, and the high-level evidence for advanced gastric cancer based on large prospective randomized controlled trial as CLASS-01、JCOG 0901, KLASS -02 is still awaited.Hopefully, it would have also gained the solid evidence of laparoscopy-assisted distal gastrectomy for the treatment of advanced gastric cancer (AGC).
* China has entered the aging society since 1999. Among the GC patients in China, the average age is 65 years old, which makes increasing attempts to explore laparoscopic techniques in the treatment of elderly patients.
* Nowadays, a considerable proportion of elderly patients suffer from multiple diseases, such as hypertension, diabetes, coronary heart disease. Thus the risk of intraoperative and postoperative complications can not be ignored. Unfortunately, there are rare studies specializing into the LAG for the GC patients of > 65 years old.
* Accordingly, the comparison of intraoperative and postoperative complications between laparoscopy-assisted and open distal gastrectomy for over 65 years old patients with gastric cancer based on a randomized controlled trial is warranted.

ELIGIBILITY:
Inclusion Criteria:

* Age over 65 years
* Primary gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by endoscopic biopsy
* cT1-4a, N0-3, M0 at preoperative evaluation according to the AJCC Cancer Staging Manual Seventh Edition
* Expected curative resection through distal subtotal gastrectomy with D2 lymphadenectomy
* Performance status of 0 or 1 on ECOG (Eastern Cooperative Oncology Group) scale
* ASA (American Society of Anesthesiology) score class I, II, or III
* Written informed consent

Exclusion Criteria:

* Severe mental disorder
* History of previous upper abdominal surgery (except laparoscopic cholecystectomy)
* History of previous gastrectomy, endoscopic mucosal resection or endoscopic submucosal dissection
* Exclude the early gastric cancer feasible for ESD
* Enlarged or bulky regional lymph node diameter over 3cm by preoperative imaging
* History of other malignant disease within past five years
* History of previous neoadjuvant chemotherapy or radiotherapy
* History of unstable angina or myocardial infarction within past six months
* History of cerebrovascular accident within past six months
* History of continuous systematic administration of corticosteroids within one month
* Requirement of simultaneous surgery for other disease
* Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer
* FEV1<50% of predicted values

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative complication rate | 30 days
  30 day morbidity and mortality

SECONDARY OUTCOMES:
Postoperative pulmonary complications | 30 days
  Pulmonary complications after operation within 30 days
Postoperative recovery index | 7 days
  participants will be followed for the duration of hospital stay after operation, an expected average of 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Guoxin Li, M.D., Ph.D., Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, China

REFERENCES:
- [Background] Yu J, Hu J, Huang C, Ying M, Peng X, Wei H, Jiang Z, Du X, Liu Z, Liu H, Li G; Chinese Laparoscopic Gastrointestinal Surgery Study (CLASS) Group. The impact of age and comorbidity on postoperative complications in patients with advanced gastric cancer after laparoscopic D2 gastrectomy: results from the Chinese laparoscropic gastrointestinal surgery study (CLASS) group. Eur J Surg Oncol. 2013 Oct;39(10):1144-9. doi: 10.1016/j.ejso.2013.06.021. Epub 2013 Jul 10. PMID 23850088
- [Derived] Luo J, Zhu Y, Liu H, Hu YF, Li TJ, Lin T, Chen T, Chen H, Chen XH, Yu J, Li GX. Morbidity and mortality of elderly patients with advanced gastric cancer after laparoscopy-assisted or open distal gastrectomy: a randomized-controlled trial. Gastroenterol Rep (Oxf). 2018 Nov;6(4):317-319. doi: 10.1093/gastro/goy013. Epub 2018 May 17. PMID 30430021
- See also: Southern Medical University, China — http://www.fimmu.com/index_com.html
- See also: Nanfang Hospital, China — http://www.nfyy.com/
- See also: Chinese Anti-Cancer Association — http://www.caca.org.cn/